CLINICAL TRIAL: NCT03637803
Title: A Phase I/II Open Label, Safety And Preliminary Efficacy Study of MRx0518 In Combination With Pembrolizumab In Patients With Advanced Malignancies Who Have Progressed On PD-1/PD-L1 Inhibitors
Brief Title: Live Biotherapeutic Product MRx0518 and Pembrolizumab Combination Study in Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor insolvency
Sponsor: 4D pharma plc (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRx0518-I-002; Keynote MK3475-823 (Other: Merck)
Record Dates: First submitted 2018-08-03; First posted 2018-08-20 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Oncology; Solid Tumor; Non Small Cell Lung Cancer; Renal Cell Carcinoma; Melanoma; Bladder Cancer
Keywords: MK-3475; pembrolizumab; MRx0518; PD-1 Inhibitor; Oncology; Live Biotherapeutic Product
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Melanoma; Urinary Bladder Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MRx0518 with pembrolizumab (Experimental): Subjects will receive IV infusion of pembrolizumab once every 3 weeks until disease progression, unacceptable AEs or withdrawal of consent up to a maximum of 35 cycles (approx. 2 years). Starting on the day of first pembrolizumab dose, subjects will take one capsule of MR0518 twice daily until the end of the treatment period.
  Interventions: Drug: MRx0518; Drug: Pembrolizumab 25 MG/1 ML Intravenous Solution [KEYTRUDA]

INTERVENTIONS:
Drug: MRx0518 — MRx0518 is a live biotherapeutic product consisting of a lyophilised formulation of a proprietary strain of bacterium. The study dosing regimen is one capsule two times per day for the duration of the treatment period.
Drug: Pembrolizumab 25 MG/1 ML Intravenous Solution [KEYTRUDA] — Pembrolizumab is a potent humanised immunoglobulin G4 (IgG4) monoclonal antibody (mAb) with high specificity of binding to the programmed cell death 1 (PD1) receptor , thus inhibiting its interaction with programmed cell death ligand 1 (PD-L1) and programmed cell death ligand 2 (PD-L2). The study dosing regimen is 200mg (two 4ml vials of 25mg/ml solution) for IV infusion once every three weeks.
  Other Names: MK3475; Pembrolizumab; Keytruda

SUMMARY:
This is an open label, safety and preliminary efficacy study of MRx0518 in combination with pembrolizumab in patients with solid tumours (non small cell lung cancer, renal cell carcinoma, bladder cancer or melanoma).

Subjects will be treated with IV pembrolizumab every 3 weeks and 1 capsule twice daily of MRx0518. Treatment will continue as long as clinically relevant, until disease progression, unacceptable AEs or withdrawal of consent up to a maximum of 35 cycles (approx. 2 years).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent/assent for the trial.
* ≥18 years of age on day of signing informed consent.
* Histological or cytological evidence of advanced and/or metastatic or recurrent NSCLC, renal cell carcinoma, bladder cancer or melanoma.
* At least one measurable lesion per RECIST v 1.1 criteria.
* Failure to respond or intolerance to standard therapy or for whom no appropriate therapies are known to provide clinical benefit (per the judgement of the Investigator).
* Subjects must have progressed on treatment with a PD-1/PD-L1 inhibitor administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies. PD-1/PD-L1 inhibitor treatment progression is defined by meeting all of the following criteria:

  1. Has received at least 2 doses of a PD-1/PD-L1 inhibitor.
  2. Has demonstrated disease progression after PD-1/PD-L1 therapy as defined by RECIST v1.1, iRECIST or irRECIST. The initial evidence of disease progression (PD) is to be confirmed by a second assessment no less than four weeks from the date of the first documented PD, in the absence of rapid clinical progression.
  3. Progressive disease has been documented within 12 weeks from the last dose of a PD-1/PD-L1 inhibitor.
* Have adequate organ function
* Be willing to provide archival tissue
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Female subjects of childbearing potential should have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for ≥2 years.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication
* Male subjects with female partners of childbearing potential should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Subjects who failed to show any response to initial treatment with PD-1/PD-L1 inhibitor (i.e. no Response or no Stable Disease).
* Has active brain metastases or leptomeningeal disease. Subjects with asymptomatic CNS metastases which have been stable (defined as without evidence of progression by MRI for at least 28 days prior to initiation of therapy and any neurologic symptoms have returned to baseline) following treatment with surgery or radiation therapy are allowed.
* Prior solid organ or hematologic transplant.
* Treatment-related immune-mediated (or immune related) AEs from immune-modulatory agents (including but not limited to anti-PD1/PD-L1 agents, anti-CTLA4 monoclonal antibodies) that caused permanent discontinuation of the agent, or that were grade 3 or 4 in severity.
* Subjects treated with chemotherapy, immunotherapy, biologic therapy, or other investigational agent within <5 times the half-life of the agent or <21 days (whichever is shorter) of starting study drug. Continuation of hormone replacement therapy is permitted. Stable regimens of hormonal therapy i.e. for prostate cancer (e.g. leuprolide, a GnRH agonist), ovarian, or breast cancer are not exclusionary.
* Subjects treated with tyrosine kinase inhibitor therapy or completed palliative radiotherapy <14 days from initiation of therapy.
* Comorbidity requiring corticosteroid therapy (>10mg prednisone/day or equivalent) within 7 days of starting experimental therapy. Physiologic replacement doses are allowed if they are ≤10mg of prednisone/day or equivalent, as long as they are not being administered for immunosuppressive intent. Inhaled or topical steroids are permitted, provided that they are not for treatment of an autoimmune disorder.
* Significant cardiac dysfunction, New York Heart Association classification for chronic heart failure III-IV, symptomatic coronary artery disease, significant ventricular arrhythmias; myocardial infarction within 6 months; unstable, poorly controlled angina pectoris
* Active, known or suspected autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs), except for replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.). Note: corticosteroids given within 24 hours of an imaging study for purposes of pre-medication in subjects with hypersensitivity to radiologic contrast agents are allowed
* Has a serious active infection requiring systemic therapy
* Subjects who have completed a course of antibiotics within the two weeks prior to dosing
* Has a known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the trial
* Receipt of a live-virus vaccination within 28 days of planned treatment start
* Known HIV infection, or active infection with hepatitis A, B or C
* Has a history of (non-infectious) pneumonitis that required steroids or has current active pneumonitis
* Known additional malignancy either progressing r requiring active treatment (except for non-melanoma skin cancer, in situ cervical cancer or prostate intraepithelial neoplasia) within the last 2 years
* Female subjects who are breastfeeding
* Known intolerance or hypersensitivity to study drugs
* Subjects who are allergic to amoxicillin/clavulanic acid, erythromycin and imipenem
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has a known inability for oral intake of capsules

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Part A: To assess the safety and tolerability of MRx0518 in combination with pembrolizumab through the collection of adverse events | Baseline to treatment discontinuation up to a maximum of 35 treatment cycles (one cycle = 21 days)
  Adverse events will be assessed as per CTCAE v4
Part B: To assess safety and tolerability of MRx0518 in combination with pembrolizumab through the collection of adverse events | Baseline to treatment discontinuation up to a maximum of 35 treatment cycles (one cycle = 21 days)
  Adverse events will be assessed as per CTCAE v4
Part B: To assess the clinical benefit of MRx0518 in combination with pembrolizumab | Baseline to treatment discontinuation up to a maximum of 35 treatment cycles (one cycle = 21 days)
  To determine preliminary evidence of anti-tumor activity

SECONDARY OUTCOMES:
Antitumour effect | Baseline and every 3 weeks until treatment discontinuation up to a maximum of 35 treatment cycles (one cycle = 21 days)
  Antitumour effect is assessed through tumour imaging and measurement of lesions per RECIST and iRECIST (ORR, DOR, DCR, PFS)

OTHER OUTCOMES:
Biomarkers of treatment effect - blood | Day 1 of Cycle 1 and Cycle 2 and time of treatment discontinuation up to a maximum of 35 treatment cycles (one cycle = 21 days)
  Blood samples will be analysed for changes in immune status and biomarkers of treatment effect
Biomarkers of treatment effect - tumour | Baseline, Day 1 of Cycle 4 and time of treatment discontinuation up to a maximum of 35 treatment cycles (one cycle = 21 days)
  Tissue biopsies will be taken to analyse for tumour biomarkers
Microbiota and metabolome | Day 1 of Cycle 1 and Cycle 2, time of treatment discontinuation up to a maximum of 35 treatment cycles (one cycle = 21 days), and 30 Day follow up
  Faecal and urine samples will be collected and analysed for microbiota and metabolomics using the MicroDx platform
Overall survival | From start of treatment until death due to any cause up to a maximum of 35 treatment cycles (one cycle = 21 days)
  Survival of the subjects will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Shubham Pant, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - University of Kansas Medical Center, Kansas City, Kansas
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Houston Methodist Cancer Center, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Summit Cancer Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No